CLINICAL TRIAL: NCT04551443
Title: Randomised, Double-blind, Placebo-controlled, Intravenous Infusion Human Wharton' Jelly-derived Mesenchymal Stem Cells in Patients With Acute Myocardial Infarction
Brief Title: WJMSCs Anti-inflammatory Therapy in Acute Myocardial Infarction
Acronym: WAIAMI
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Navy General Hospital, Beijing (Other)
Collaborators: Peking University Third Hospital (Other); Peking Union Medical College Hospital (Other); Xijing Hospital (Other); Chinese PLA General Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PLAG6C
Record Dates: First submitted 2019-12-12; First posted 2020-09-16 (Actual); Last update posted 2020-09-16 (Actual); Status verified 2019-12

CONDITIONS: Acute Myocardial Infarction
Keywords: AMI;; Mesenchymal Stem Cells;; anti-inflammatory;

STUDY DESIGN:
Intervention Model Description: Placebo Comparator: Intravenous infusion WJMSCs +standard therapy Vs placebo+ standard therapy in patients with acute myocardial infarction
Who Masked: Participant, Investigator
Masking Description: The eligible patients were assigned randomly to each of two groups (WJMSCs or placebo control) in a 1:1 fashion using a computer-generated randomization of sequence numbers. Physicians and other clinical personnel remained blind to the treatment assignment throughout the study.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Placebo PBS (Placebo Comparator): Standard therapy+Intravenous infusion PBS in patients with AMI
  Interventions: Biological: Intravenous infusion placebo; Biological: Intravenous infusion WJMSCs
- WJMScs (Active Comparator): Standard therapy+Intravenous infusion WJMSCs in patients with AMI
  Interventions: Biological: Intravenous infusion placebo; Biological: Intravenous infusion WJMSCs

INTERVENTIONS:
Biological: Intravenous infusion placebo — Intravenous infusion placebo or WJMSCs in patients with AMI
  Other Names: PBS
Biological: Intravenous infusion WJMSCs — Intravenous infusion WJMSCs or placebo in patients with AMI
  Other Names: WJMSCs

SUMMARY:
Cumulative evidence has demonstrated that cardiac repair after acute myocardial infarction (AMI) is characterized by a series of time-dependent events orchestrated by the innate immune system. This begins immediately after the onset of necrotic cell death with intense sterile inflammation and myocardial infiltration of a variety of immune cell subtypes including monocytes and macrophages during the first several days after MI. There is increasing evidence to suggest inflammation is not limited to the infarcted myocardium and systemic imbalances in the post-infarct inflammatory cascade can exacerbate adverse remodelling beyond the infarct site. Therefore, it is very important that therapies seek to target the intricate balance between pro- and antiinflammatory pathways timely after AMI. Human mesenchymal stem cells (hMSCs) have been shown to exhibit immunomodulation, angiogenesis, and paracrine secretion of bioactive factors that can attenuate inflammation and promote tissue regeneration, making them a promising cell source for AMI therapy. However, it has been proved in our and other studies that perfusion of WJMSCs after 5 days of AMI can only slightly improve left ventricular end-diastolic volume, which is the most important indicator of left ventricular remodeling. Thus, WANIAMI Trial is a randomized, double-blind, placebo controlled, phase#study designed to assess the safety and feasibility of intravenous infusion of WJMSCs in the treatment of patients in the acute phase ( within 24h) with the both of ST-Segment-Elevation or Non-ST-Segment-Elevation AMI.

DETAILED DESCRIPTION:
At present, although the implementation of timely reperfusion strategies has reduced the acute mortality associated with AMI, improved patient survival has increased the incidence of chronic heart failure, due in large part to adverse remodeling of the damaged left ventricle (LV) following the initial ischemic event. However, recently, pathophysiological mechanisms of AMI reveal that begins immediately after the onset of necrotic cell death with intense sterile inflammation and myocardial infiltration of a variety of immune cell subtypes including neutrophils, monocytes and macrophages during the first several days after MI. Improved understanding in the interactions between cells, extracellular matrix (ECM) and signaling molecules within the injured myocardium have allowed development of novel experimental therapies. These therapies seek to target the intricate balance between pro- and anti-inflammatory pathways in an attempt to limit ischemic injury and prevent subsequent development of heart failure. Mesenchymal stem cells (MSCs), in particular, have emerged as potent paracrine modulators of inflammation that promote myocardial healing after infarction.

The latest cell biological studies have demonstrated that mesenchymal stem cells have a unique immunomodulatory function. MSCs contribute to a critical role in regulating the inflammatory microenvironment and interacting with immune cells, including T cells, B cells, natural killer (NK) cells, and dendritic cells (DCs). MSC induce anti- inflammatory macrophages, inhibit foam cell formation, suppress immune responses of endothelial cells and innate lymphoid cells, and increase phagocytic capacity, which indirectly suppresses T cell proliferation. In mouse AMI models, we found MSCs transplantation significantly reduced the number of inflammatory macrophages (M1), increased the number of anti-inflammatory macrophages (M2) and prevented the expansion of AMI during early stage of AMI. More recently, the paracrine potency might vary with sources and microenvironment of MSCs. MSCs isolated from fetal tissues such as umbilical cord (UC) and UC-blood (UCB) were shown to have increased secretion of anti-inflammatory factors (TGF-β,IL-10) and growth factors than MSCs obtained from adult adipose tissue or bone marrow. Our previous research found that the expression characteristics of special immunomodulatory genes of human umbilical cord Wharton's jelly-derived MSCs (WJMSCs). At present, many studies have demonstrated WJMSC possess s a robust immunomodulatory potential and anti-inflammatory effects through release of secretome consisting of a diverse range of cytokines, chemokines, and extracellular vesicles (EVs), the cross talk and interplay of WJMSCs and local environment reversely control and regulate the paracrine activity of MSCs. Thus WJMSCs are important regulators of immune responses and may hold great potential to be used as a therapeutic in AMI. In particular#safety and feasibility of WJMSCs transplant have been clearly proved by us and other studies in patients with AMI.

Given the current evidence, systemic paracrinemediated anti-inflammatory effects of WJMSCs can drive beneficial in therapy of AMI. These concepts lead to a potentially transformative strategy that intravenous delivery of WJMSCs, through systemic anti-infammatory mechanisms.

Therefore, the investigators performed a double-blind, placebo- controlled trial, randomly assigning 200 patients with AMI to receive three times at 30-day intervals for equal doses of 1x106 /kg of WJMSCs, first time infusing within 24h after AMI or placebo , to investigate the therapeutic efficacy and safety of WJMSCs in patients with acute ST-Segment-Elevation or Non-ST-Segment-elevation myocardial infarction.

ELIGIBILITY:
Inclusion Criteria:

* Age limited ≥ 18 years at Visit 1
* Patient must provide written informed consent
* Have a diagnosis of acute ST-Segment-Elevation or Non-ST-Segment-Elevation myocardial infarction as defined by any of the following criteria:
* According to the Third Universal Definition of Myocardial Infarction Type:

Type 1 spontaneous myocardial infarction Type 2 myocardial infarction secondary to an ischemic imbalance Type 3 myocardial infarction resulting in death when biomarker values are unavailable Including: acute ST-Segment-Elevation or Non-ST-Segment-Elevation myocardial infarction, creatine kinase (CK)-MB levels over three-fold the upper limit of the reference values.

* Successful or unsuccessful. revascularization by percutaneous coronary intervention, within 12 hours after symptom onset with stent implantation and thrombolysis.

Exclusion Criteria:

* Myocardial infarction related to stent thrombosis; Myocardial infarction related to restenosis
* Myocardial infarction related to coronary artery bypass grafting (CABG)
* Have a hematologic abnormality as evidenced by hematocrit <25% , white blood cell <2500/u L or platelet values<100000/u L without another explanation.
* Have liver dysfunction , as evidenced by enzymes (aspartate aminotransferase and alanine aminotransferase) >3× the upper limits of normal
* Have a coagulopathy (international normalized ratio > 1.3) not because of a reversible cause (ie, coumadin)
* Be an organ transplant recipient
* Have a clinical history of malignancy within 5 y except curatively treated basal cell carcinoma, squamous cell carcinoma, or cervical carcinoma.
* Have a noncardiac condition that limits lifespan to <1y.
* Have a history of drug or alcohol abuse within the past 24 m.
* Be serum positive for human immunodeficiency virus, hepatitis B surface antigen, or hepatitis C.
* Be a female who is pregnant, nursing, or of childbearing potential who is not practicing effective contraceptive methods.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2020-11-01 (Estimated); Primary Completion 2021-12-30 (Estimated); Study Completion 2022-12-30 (Estimated)

PRIMARY OUTCOMES:
Any composite of major adverse cardiovascular events | 12 months
  The main safety endpoints was the first occurrence of a major adverse cardiovascular event (a composite of nonfatal myocardial infarction, nonfatal stroke, or cardiovascular death) and hospitalization for unstable angina that led to urgent coronary revascularization within 12 months.
Checking patient LVEF | 6 months
  The main feasibility endpoints were defined as the change in LVEF, infarct size as determined by MRI and perfusion defect as assessed by MIBI SPECT from baseline to 6 months.
Checking patient infarct size | 6 months
  The main feasibility endpoints were defined as the change in infarct size
checking patient perfusion defect. | 6 months
  The main feasibility endpoints were defined as non significant perfusion defect

SECONDARY OUTCOMES:
Coronary disease | 12 months
  Secondary end points included death from a composite of major adverse card cardiovascular events plus any coronary revascularization within 12 months.
Coronary congestive heart failure | 12 months
  Secondary end points included death from hospitalization for congestive heart failure within 12 months.
Coronary changes in hsCRP | 12 months
  Secondary end points included the level change of hsCRP within 12 months.

CONTACTS AND LOCATIONS:
Overall Officials: Lian Ru Gao, MD, Study Chair — The Sixth Medical Center of P.L.A. General Hospital

IPD SHARING:
Plan to Share IPD: Undecided